CLINICAL TRIAL: NCT05459324
Title: Effects of Novel SCS Paddle on Intraoperative Neuromonitoring Recording: Phase II
Brief Title: Intraoperative Neuromonitoring Recording With a Novel SCS Paddle: Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 6426 Microleads
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain; Neuropathic Pain; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes
Keywords: Spinal cord stimulation; chronic pain
MeSH Terms: conditions — Chronic Pain; Neuralgia; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Statistics will be performed comparing the HR-SCS to commercial SCS devices. Additionally, we will correlate patient reported outcomes and spinal measurements to IONM outcomes to determine overall device capabilities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study Group (Experimental): Twenty-four patients offered SCS for standard of care were also invited to participate in this study, in which a study electrode was temporarily placed intraoperatively and neuromonitoring was done per our routine standard-of-care
  Interventions: Device: HD Study Electrode

INTERVENTIONS:
Device: HD Study Electrode — The HD Study Electrode is an array of 8 columns of stimulation contacts arranged in 8 rows with a low-volume electrode body. This array of stimulation electrodes contact patterns of bi-poles and tri-poles may be applied to the spinal cord for assessment of dermatomal selective stimulation patterns.

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of a new spinal cord stimulation paddle electrode which is able to target the dorsal horns, dorsal nerve roots, and dorsal columns. The research electrode ("Study Electrode") is designed to answer basic physiological clinical research questions. It may inform future device therapy development, but the Study Electrode is not a product that will be marketed or sold. The Investigators believe the protocol is a Non-Significant Risk study answering basic physiological research questions, which may be performed under hospital IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a spinal cord stimulation procedure for neuropathic pain.
* have undergone a successful SCS trial and are determined eligible for a permanent SCS implant.
* Patients must be fluent in English as well as mentally competent to read and answer the questionnaires, as well as complete pain assessment exams.-
* subjects must be able to give informed consent.

Exclusion Criteria:

* patients who are not undergoing thoracic spinal cord stimulation for chronic neuropathic pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 3 months
  Patients rate their pain on a scale from 0-10; 0 being not in pain and 10 being worst pain imaginable. A higher score indicates worse outcome.

SECONDARY OUTCOMES:
McGill Pain Questionnaire (MPQ) | 3 month
  Patients select words that describe their pain. There are a total of 15 words. A higher score (more words selected) indicates worse outcome with a range from 0-15.
Oswestry Disability Index (ODI) | 3 months
  This is a multiple choice style scale where patients are presented with an activity and asked to select a description which best matches their ability to perform that activity. Multiple choice options are then scored on a scale from 0-5; where 0 is no issues performing the activity and 5 is cannot perform activity. A higher score indicates worse outcome. The range in scores is from 0-100.
Pain Catastrophizing Scale (PCS) | 3 months
  Patients are presented with a series of statements and they are asked to rate on a scale from 0-4, how often these statements apply to them when they are in pain. 0= never and 4= always. A higher score indicates worse outcome. Scores range from 0-52.
Beck Depression Index (BDI) | 3 months
  This is a multiple choice style scale where patients are asked to select a statement related to a feeling of sadness or a component of depression. Multiple choice options are then scored on a scale from 0-3; where 0 is they do not feel that way and 3 is they do feel that way. A higher score indicates worse outcome. Scores range from 0-63

OTHER OUTCOMES:
PainDetect | Baseline
  Ensures patient's pain is neuropathic in nature

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States

REFERENCES:
- [Derived] Berwal D, Quintero A, Telkes I, DiMarzio M, Harland T, Paniccioli S, Dalfino J, Iyassu Y, McLaughlin BL, Pilitsis JG. Improved Selectivity in Eliciting Evoked Electromyography Responses With High-Resolution Spinal Cord Stimulation. Neurosurgery. 2024 Aug 1;95(2):322-329. doi: 10.1227/neu.0000000000002878. Epub 2024 Feb 20. PMID 38376181